CLINICAL TRIAL: NCT04588584
Title: Prescribing Practice of Medicinal Products From the Perspective of the Patient.
Brief Title: Prescribing Practice of Medication - Patient View.
Status: Completed | Type: Observational
Sponsor: Medical University of Graz (Other)
Responsible Party: Sponsor
Other Study IDs: EK_NR_30-178 ex 17/18
Record Dates: First submitted 2020-10-08; First posted 2020-10-19 (Actual); Last update posted 2020-10-19 (Actual); Status verified 2020-10

CONDITIONS: Focus: Prescribing Practice
MeSH Terms: interventions — Surveys and Questionnaires; Interviews as Topic

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Survey and Interviews — Survey and Interviews

SUMMARY:
In the clinical routine of a hospital, there are often problems dealing with medication that has already been prescribed at the time of admission due to incomplete or missing medication lists from the family doctor. Often patients forget this list at home.

This pilot study focuses on the medication process from admission to discharge and patient health literacy.

ELIGIBILITY:
Inclusion Criteria:

* Patient hospitalised at the clinical ward of Endocrinilogy and Diabetology and plastic Surgery
* Patient with an minimum of 2 days hospitalisation
* good knowledge of German
* Age 18 to 99 Years
* Male/female

Exclusion Criteria:

* Neurological or psychiatric primary disease e.g. Dementia
* Rehospitalisation 7 days after discharge from hospital
* Patients who need intensive care

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 100 patients in the primary care clinic
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2018-02-19 (Actual); Primary Completion 2020-07-31 (Actual); Study Completion 2020-09-30 (Actual)

PRIMARY OUTCOMES:
Health competence of patients with focus on drugs. | 6 months
  Correct knowledge of the medication (indication) - assessed by Interview with the patient
Drug prescription from the view of the patient- Amount | 6 months
  Amount of prescribed drugs by descriptive chart review with CRF (Case Report Form) and interview with the patient
Drug prescription from the view of the patient- Type of drugs | 6 months
  Type of prescribed drugs by descriptive chart review with CRF and interview with the patient
Drug prescription from the view of the patient- Discrepancies | 6 months
  Potential discrepancies between amount or type of drugs indicated by the patient and descriptive chart review with CRF

CONTACTS AND LOCATIONS:
Locations (1):
- LKH University clinical Graz , QM-RM, Graz, Styria, Austria